CLINICAL TRIAL: NCT04678401
Title: A Pilot/Phase 1 Study of Immunosuppression-free Regulatory T-cell Graft-engineered Haploidentical Hematopoietic Cell Transplantation in Relapsed/Refractory and Ultra-High-risk AML/MDS
Brief Title: IS-free Treg HaploHCT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, John Koreth, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-336
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Stem Cell Transplant Complications; Graft Vs Host Disease; Myeloid Leukemia, Acute; Myeloid Leukemia in Relapse (Disorder); Myelodysplastic Syndromes
Keywords: Stem Cell Transplant Complications; Graft Vs Host Disease; Myeloid Leukemia, Acute; Myeloid Leukemia in Relapse (Disorder); Myelodysplastic Syndromes
MeSH Terms: conditions — Graft vs Host Disease; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Radiation; Radiotherapy; Whole-Body Irradiation; fludarabine; fludarabine phosphate; Thiotepa; Cyclophosphamide; Mesna; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IS-FREE TREG GRAFT_ENGINEERED HaploHCT for relapsed/refractory AML or MDS EB-2 (Closed to Accrual) (Experimental): Please note that this arm is closed due to meeting accrual goal as of June 2024.
  This arm (Cohort A) included patients with rel/ref AML/MDS, with active disease despite at least 1 prior line of therapy.
  Treatment plan and follow up schedule:
  Day -15 to -6: Myeloablative conditioning regimen Radiation: Total Myeloid and Lymphoid Irradiation (TMLI) on Days -15 to -11 OR Total Body Irradiation (TBI) on Days -13 to -11 Chemotherapy: Fludarabine on Days -10 to -6, Thiotepa on Days -10 to -9, and Cyclophosphamide and Mesna on Days -8 and -7
  Day -4: Treg-enriched donor cell infusion and GVHD assessment
  Day -1: Unmodified donor T Cell infusion and GVHD assessment
  Day 0: CD34+ Haplo Peripheral Blood Stem Cell Transplant and GVHD assessment
  Days 30, 60, 100, 180, 365 post-HSCT, participants will undergo testing and assessment of minimal residual disease (MRD) and (GVHD).
  Interventions: Radiation: Radiation; Drug: Fludarabine; Drug: Thiotepa; Drug: Cyclophosphamide; Drug: Mesna; Biological: Treg-enriched donor cell; Biological: Unmodified donor T Cell; Procedure: CD34+ Haplo Peripheral Blood Stem Cell
- IS-FREE TREG GRAFT_ENGINEERED HaploHCT for Ultra high-risk AML or MDS with mutated TP53 (Experimental): This arm (Cohort B) includes patients with ultra-high-risk AML/MDS that meets the definition of "Myeloid Neoplasms with mutated TP53" per the 2022 International Consensus Classification, regardless of remission status at the time of transplant.
  Treatment plan and follow up schedule:
  Day -15 to -6: Myeloablative conditioning regimen Radiation: Total Myeloid and Lymphoid Irradiation (TMLI) on Days -15 to -11 OR Total Body Irradiation (TBI) on Days -13 to -11 Chemotherapy: Fludarabine on Days -10 to -6, Thiotepa on Days -10 to -9, and Cyclophosphamide and Mesna on Days -8 and -7
  Day -4: Treg-enriched donor cell infusion and GVHD assessment
  Day -1: Unmodified donor T Cell infusion and GVHD assessment
  Day 0: CD34+ Haplo Peripheral Blood Stem Cell Transplant and GVHD assessment
  Days 30, 60, 100, 180, 365 post-HSCT, participants will undergo testing and assessment of minimal residual disease (MRD) and (GVHD).
  Interventions: Radiation: Radiation; Drug: Fludarabine; Drug: Thiotepa; Drug: Cyclophosphamide; Drug: Mesna; Biological: Treg-enriched donor cell; Biological: Unmodified donor T Cell; Procedure: CD34+ Haplo Peripheral Blood Stem Cell
- IS-FREE TREG GRAFT_ENGINEERED HaploHCT for Ultra high-risk AML or MDS with multi-hit or CK+ mut-TP53 (Experimental): This arm (Cohort C) includes patients with ultra-high-risk AML/MDS that meets definition of 'Myeloid Neoplasms with multi-hit or complex karyotype (CK+) mutated TP53' per 2022 International Consensus Classification, with response (AML with <5% BM blasts/MDS with <10% BM blasts).
  Treatment plan and follow up schedule:
  Day -11 to -5: Reduced intensity conditioning regimen Chemotherapy: Thiotepa on Day -11, Fludarabine on Days -10 to -7, and Melphalan on Day -6 Radiation: Total Body Irradiation (TBI) on Day -5
  Day -4: Treg-enriched donor cell infusion and GVHD assessment
  Day -1: Unmodified donor T Cell infusion and GVHD assessment
  Day 0: CD34+ Haplo Peripheral Blood Stem Cell Transplant and GVHD assessment
  Days 30, 60, 100, 180, 365 post-HSCT, participants will undergo testing and assessment of minimal residual disease (MRD) and (GVHD).
  Interventions: Radiation: Radiation; Drug: Fludarabine; Drug: Thiotepa; Biological: Treg-enriched donor cell; Biological: Unmodified donor T Cell; Procedure: CD34+ Haplo Peripheral Blood Stem Cell; Drug: Melphalan

INTERVENTIONS:
Radiation: Radiation — For MAC regimen:
  Total Myeloid and Lymphoid Irradiation (TMLI) delivered through Radiation Oncology institutional standards and comprised of 13.5 Gy TMI (9 fractions, 1.5 Gy per fraction, 2 fractions per day) and 11.7 Gy TLI (9 fractions, 1.3 Gy per fraction, 2 fractions per day).
  OR Total Body Irradiation (TBI) comprised of 12 Gy (6 fractions, 2 Gy per fraction, 2 fractions per day)
  For RIC regimen:
  TBI comprised of 2 Gy in 1 fraction.
  Other Names: Radiotherapy, TMLI, TBI
Drug: Fludarabine — For MAC regimen: 30 mg/m^2/d in 100 ml normal saline (NS) will be administered as a bolus infusion administered by IV infusion over approximately 30 minutes for 5 days (on day -10, -9, -8, -7, -6)
  For RIC regimen: 40 mg/m^2/d in 100 ml NS will be administered as a bolus by IV infusion over approximately 30 minutes for 4 days (on day -10, -9, -8, -7)
  Other Names: Fludara
Drug: Thiotepa — For MAC regimen: 3.75 mg/kg diluted in NS to a final concentration of 1mg/mL will be administered by IV infusion over approximately 4 hours daily for 2 days (on day -10, -9)
  For RIC regimen: 5 mg/kg diluted in NS to a final concentration of 1mg/mL will be administered by IV infusion over approximately 4 hours twice daily for 1 day (on day -11)
  Other Names: Tepadina
Drug: Cyclophosphamide — For MAC regimen only: 15 mg/kg diluted in NS per institutional standard and will be administered by IV over 1 hour or as directed per institutional standard practice, daily on D-8, -7.
  Other Names: cytophosphane
  Arms: IS-FREE TREG GRAFT_ENGINEERED HaploHCT for Ultra high-risk AML or MDS with mutated TP53; IS-FREE TREG GRAFT_ENGINEERED HaploHCT for relapsed/refractory AML or MDS EB-2 (Closed to Accrual)
Drug: Mesna — For MAC regimen only: 3.75mg/kg (25% of cyclophosphamide dose) diluted in 50 mL NS and administered IV over 30 min, will be infused starting 30 min prior to cyclophosphamide and for 3 doses thereafter, at 3, 6 and 9h after cyclophosphamide
  Other Names: Mesnex
  Arms: IS-FREE TREG GRAFT_ENGINEERED HaploHCT for Ultra high-risk AML or MDS with mutated TP53; IS-FREE TREG GRAFT_ENGINEERED HaploHCT for relapsed/refractory AML or MDS EB-2 (Closed to Accrual)
Biological: Treg-enriched donor cell — Target 'Treg-enriched' cell dose is 1-2 x 10^6 cells/kg. Cells will be given intravenously on Day -4. The day -1 calculated unmodified PBMC T ('Teff') cell dose will be adjusted to maintain a targeted cell ratio of 2 'Treg-enriched' cells:1 'Teff' cell.
Biological: Unmodified donor T Cell — Unmodified donor PBMCs will be infused at a calculated 'Teff' dose of 1x10^6 CD3+ T cells/kg, adjusted per the caveats below:
  A) If the 'Treg-enriched' product infused was at target dose of 2x106 cells/kg but had ≥30% CD4+CD25+CD127hi cells, the unmodified 'Teff' (calculated) cell dose infused on day -1 will be halved to 0.5x10^6 CD3+ T cells/kg.
  B) If the 'Treg-enriched' product was in the range of 1-2x106 cells/kg, the unmodified 'Teff' (calculated) cell dose on day -1 will be adjusted to between 0.5-1x10^6 CD3+ T cells/kg, dosed to maintain a 2 'Treg-enriched':1 'Teff' (calculated) ratio of infused cells.
  C) If the 'Treg-enriched' product infused met both caveats A and B above, the unmodified 'Teff' (calculated) cell dose infused on day -1 will be halved to 0.5x10^6 CD3+ T cells/kg.
Procedure: CD34+ Haplo Peripheral Blood Stem Cell — The megadose donor CD34+ PBSC infusion target is >10x10^6 CD34+ cells/kg (ABW or IBW, whichever is greater). If the CD34+ graft has <6x10^6 CD34+ cells/kg (ABW or IBW, whichever is greater) (below megadose minimum) it WILL be infused in order to rescue recipient hematopoiesis, and the patient will remain on study.
Drug: Melphalan — For RIC regimen only: 100 mg/m2 will be administered as a bolus by IV infusion over approximately 30 minutes for 1 day (on day -6)
  Other Names: Alkeran
  Arms: IS-FREE TREG GRAFT_ENGINEERED HaploHCT for Ultra high-risk AML or MDS with multi-hit or CK+ mut-TP53

SUMMARY:
This research study is evaluating the safety and efficacy of the IS-free Treg-cell graft-engineered haplo transplant method in people with relapsed/refractory and Ultra-high risk acute myeloid leukemia (AML) and/or myelodysplastic syndromes (MDS) receiving a haploidentical donor allogeneic hematopoietic stem cell transplant (HSCT).

The names of the study interventions involved in this study are:

* Radiation-Total Myeloid and Lymphoid Irradiation (TMLI)
* Chemotherapy (Fludarabine, Thiotepa, Cyclophosphamide plus Mesna)
* Infusion of haplo Treg-enriched donor cells (experimental therapy)
* Infusion of unmodified haplo donor T cells (includes cancer-fighting T effector cells)
* Infusion of haplo donor CD34+ Peripheral Blood Stem Cells

DETAILED DESCRIPTION:
This study is assessing whether the IS-free Treg-cell graft-engineered haplo HSCT approach will reduce risk of relapse while preventing usual toxicities related to stem cell transplants (e.g., graft-versus-host-disease (GVHD)).

GVHD is a complication of transplantation where the T cells (a type of white blood cell that helps protect the body from relapse by killing cancer cells) in the donor graft attack and damage some of the host tissues. Patients who receive an allogeneic (using another person as the donor) hematopoietic stem cell transplant (HSCT) may develop graft-versus-host disease (GVHD) toxicity and are also at risk of disease relapse.

The research study procedures include the following: screening for eligibility, study treatment, and follow up visits.

Participants will receive the study intervention Treg-enriched donor cells and will then be followed for 1 year after transplantation.

It is expected that about 30 people will take part in this research study.

Dana-Farber Cancer Institute research funds along with charitable donations are supporting this research study. Regeneron Pharmaceuticals, Inc. (a pharmaceutical company) supported this research study by providing funding and support for correlative laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A: Histologically confirmed disease in the prior 4 weeks, despite at least 1 prior line of therapy (e.g., 3+7 chemotherapy, HMA therapy): Rel/ref AML (de novo or secondary) with ≥5% blasts in BM (or extramedullary sites); MDS EB-2 (BM ≥10% blasts, PB 5-19% blasts).
* Cohort B: Ultra high-risk AML or MDS that meets definition of 'Myeloid Neoplasms with mutated TP53' per 2022 International Consensus Classification (Appendix L) regardless of response
* Cohort C: Ultra high-risk AML or MDS that meets definition of 'Myeloid Neoplasms with multi-hit or complex karyotype (CK+) mutated TP53' per 2022 International Consensus Classification (Appendix L) with response: AML (de novo or secondary) with <5% blasts in BM; MDS with <10% blasts in BM or PB.
* Available haploidentical HLA-matched (-A, -B, -C, -DRB1) related donor aged 18-65 years.
* Age ≥18 to 65 years for Cohort A and B. Age ≥18 to 75 years for Cohort C. Because no dosing or adverse event data are currently available on the use of IS-free haploHCT in participants <18 years of age, children are excluded from this study but will be eligible for future pediatric trials.
* ECOG performance status ≤2 (Karnofsky ≥60, see Appendix A).
* Adequate organ and marrow function as defined below:

  * Pulmonary Function: FEV1, FVC and DLCO ≥ 60% of predicted (corrected for hemoglobin)
  * Cardiac Ejection Fraction ≥ 45%, and no evidence of pulmonary hypertension
  * Hepatic: Total bilirubin within normal institutional limits (exception permitted in Gilbert's Syndrome after discussion with study PI, on a case-by-case basis); and AST (SGOT)/ALT (SGPT) <2x institutional upper limit of normal
  * Renal: Serum Creatinine within normal institutional limits or creatinine clearance >50 mL/min/1.73 m2 (see Appendix B) for participants with creatinine levels above institutional normal.
* The effects of IS-free haploHCT on the developing human fetus are unknown. For this reason and because radiation and chemotherapeutic agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and a minimum of 4 months after completion of study.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had cytotoxic chemotherapy or radiotherapy within 2 weeks (4 weeks for nitrosoureas or mitomycin C) prior to entering the study. Use of hydroxyurea, HMA, e.g., azacytidine, decitabine) and/or FDA-approved novel targeted agents (e.g., venetoclax, FLT-3 inhibitors, IDH 1/2 inhibitors) are permitted up to a day prior to start of HCT conditioning.
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual non-hematologic toxicities > Grade 1) with exception of alopecia, unless cleared by study PI.
* Participants who received Mylotarg or other therapies associated with increased risk of hepatic veno-occlusive disease (VOD) or have known prior or active VOD. All novel therapies will be reviewed with PI.
* Participants who are receiving any other investigational agents within 21 days (or 5 half-lives) prior to study entry, whichever is longer, unless cleared by the study PI.
* Participants with extramedullary disease at immune privileged sites (e.g., CNS, testes, eye) are excluded, as these sites are less susceptible to the curative graft vs. leukemia effect of HCT.
* Myocardial infarction within 2 years prior to enrollment.
* Venous thromboembolic event (VTE) of DVT/ PE within 1 year prior to enrollment, unless approved by study PI. Patients with line-associated DVT within the past year may be enrolled if they have completed anticoagulation therapy.
* Stroke or transient ischemic attack (TIA) within 1 year prior to enrollment.
* History of bleeding peptic ulcer disease, erosive gastritis, intestinal perforation or clinically significant gastrointestinal (GI) hemorrhage or hemoptysis within the prior 6 months.
* Patients with a history of thrombotic microangiopathy (TMA) or hemolytic uremic syndrome/thrombotic thrombocytopenic purpura (HUS/TTP).
* History of life-threatening reactions to iron infusions or murine antibody-containing products.
* Known donor-specific antibodies (DSA) in the recipient of clinical significance (e.g., requiring DSA depletion with plasmapheresis, rituximab) are excluded.
* Inability to withhold agents that may interact with hepatic cytochrome P450 enzymes involved in cyclophosphamide and/or thiotepa metabolism (see Section 5.5) during day -10 through day -5. It is acceptable use alternative non-interacting medications during this period, and then restart prior medications
* Participants with uncontrolled bacterial, viral or fungal infections (i.e., currently taking medications with progression of clinical symptoms or signs).
* Recipients of prior allogeneic or autologous hematopoietic cell transplantation, or solid organ transplantation.
* Prior radiation exposure or other medical condition (e.g., Fanconi syndrome) that precludes use of myeloablative radiation (TMLI).
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with the multiple agents used routinely in myeloablative allogeneic stem cell transplantation. In addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Participants seropositive for hepatitis B or C infection are ineligible as they are at high risk of lethal treatment-related hepatotoxicity after myeloablative HCT.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because radiation and conditioning chemotherapy has the potential for teratogenic or abortifacient effects. A negative pregnancy test is required for females of childbearing potential. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with IS-free haploHCT breastfeeding should be discontinued if the mother is treated with IS-free haploHCT.
* Participants with a history of another non-hematologic malignancy are ineligible except for the following circumstances: Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | 30 days after hematopoietic cell transplantation (HCT)
  Safety will be assessed by dose-limiting toxicities (DLT) summarized by patient, type and grade as defined by the CTCAE v5.0.

SECONDARY OUTCOMES:
Engraftment rate | 30 days after hematopoietic cell transplantation (HCT)
  Will be summarized descriptively and estimated in the competing risks framework treating death without GVHD or without engraftment as a competing event depending on the actual enrolled and evaluable number of patients.
secondary graft failure rate | 100 days after hematopoietic cell transplantation (HCT)
  Will be summarized descriptively and estimated in the competing risks framework treating death without GVHD or without engraftment as a competing event depending on the actual enrolled and evaluable number of patients.
graft vs host disease (GVHD) Rate | 180 days after hematopoietic cell transplantation (HCT)
  Incidence of grade II-IV and III-IV acute graft vs host disease (GVHD) by day 180 after HCT
Mortality Rate-GVHD Relapse | 12 months after hematopoietic cell transplantation (HCT)
  Will also be summarized descriptively, estimated in the competing risks framework treating each event as a competing event. Corresponding 95% CIs will be provided.
Mortality Rate-GVHD Non- Relapse | 12 months after hematopoietic cell transplantation (HCT)
  Will also be summarized descriptively, estimated in the competing risks framework treating each event as a competing event. Corresponding 95% CIs will be provided.
Survival Rate-Relapse-Free | 12 months after hematopoietic cell transplantation (HCT)
  Estimated using Kaplan-Meier method with exact pointwise confidence intervals
Progression Free-Survival (PFS) | 12 months after hematopoietic cell transplantation (HCT)
  Estimated using Kaplan-Meier method with exact pointwise confidence intervals
Survival Rate-Relapse-Free-GVHD | 12 months after hematopoietic cell transplantation (HCT)
  Estimated using Kaplan-Meier method with exact pointwise confidence intervals
Overall survival rate | 12 months after hematopoietic cell transplantation (HCT)
  Estimated using Kaplan-Meier method with exact pointwise confidence intervals

CONTACTS AND LOCATIONS:
Overall Officials: John Koreth, MBBS, DPhil, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu